CLINICAL TRIAL: NCT02238574
Title: Chromosomal Instability as an Indicator for the Treatment of Progressive Mucosal Lesions of the Oral Cavity.
Brief Title: Diagnostics for the Treatment of Progressive Mucosal Lesions of the Oral Cavity: a Prospective Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL46343.068.13
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2014-09

CONDITIONS: Chromosomal Instability; Low Grade Dysplasia Oral Cavity; Loss of Heterozygostiy; Fluorescence In Situ Hybridization
MeSH Terms: conditions — Chromosomal Instability | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- follow up & surgery (Experimental): CIN positive with surgery and intensified follow up
  Interventions: Procedure: surgery; Other: follow up
- follow up (Active Comparator): CIN positive, only intensified outpatient follow up
  Interventions: Other: follow up

INTERVENTIONS:
Procedure: surgery — excision or carbondioxide laser evaporation of the mucosal lesion of the oral cavity
  Arms: follow up & surgery
Other: follow up — Intensified outpatient follow up (16 visits in 5 years)

SUMMARY:
Despite improvements in therapy, head and neck carcinomas still have a poor prognosis with a 5-year survival of ~ 50%. Malignancies of the head and neck area are (almost) always preceded by precursor lesions. Treatment of these premalignant mucosal abnormalities is generally limited and not very inconvenient for the patient. If this precursor lesion remain untreated, it may develop into a malignancy of the head and neck. Extensive treatment will be necessary. This means loss of function of the mouth, eg chewing, speaking and swallowing.

The hypothesis is that chromosomal instability (CIN) detected by fluorescence is situ hybridization (FISH) is a reliable indicator for progression to malignancy. By intensifying the follow up and treatment in premalignant CIN lesions, the incidence of progression to invasive carcinoma is expected to be significantly reduced. If this hypothesis is justified, there will be a place for CIN detection as a risk indicator in the diagnostic work up of premalignant lesions in the head and neck.

The investigators second hypothesis is that loss of heterozygosity (LOH) detected bij DNA markers is a reliable indicator for progression to malignancy. By intensifying the outpatient clinic follow up and treatment in premalignant lesions, the incidence of progression to invasive carcinoma is expected to be significantly reduced. If this hypothesis is justified, there will be a place for CIN and LOH detection as a risk indicator in the diagnostic work up of premalignant lesions in the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* subjects ≥18 years
* premalignant lesions of the oral cavity, classified as hyperkeratosis, hyperplasia, mild or moderate dysplasia
* written informed consent

Exclusion Criteria:

* former malignancy or lesion classified as severe dysplasia or carcinoma in situ at the same anatomical localization of the oral cavity
* lesions within an anatomical field which has been exposed to former treatment (e.g. radiotherapy)
* insufficient biopsy material to perform additional FISH analysis
* pregnancy, because of the physical burden (e.g. extra general anesthesia) in this study setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients (CIN negative and positive) who will show progression to malignancy of the oral cavity. | 1 year
  The primary goal of this prospective study is:
  1. Demonstrating the predictive value of the detection of CIN in premalignant lesions of the oral cavity by the use of FISH for the occurrence of progression to severe dysplasia /CIS or invasive carcinoma.
  2. The prevention of progression of premalignant lesions of the oral cavity to severe dysplasia / CIS or invasive carcinoma by the treatment of selected high-risk lesions.

SECONDARY OUTCOMES:
Number of patients (LOH negative and positive) who will show progression to malignancy of the oral cavity. | 1 year
  The secondary objective of this study is as follows:
  Demonstrating the predictive value of the detection of LOH in premalignant lesions of the oral cavity by the use of DNA markers for the occurrence of progression to severe dysplasia / CIS or invasive carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Borgemeester, MD, Study Director — University medical centre Maastricht
Locations (1):
- Maastricht Universitair Medisch Centrum (MUMC), Maastricht, Limburg, Netherlands